CLINICAL TRIAL: NCT02549274
Title: Effectiveness of Active Home Exercises for Patients With Chronic Neck Pain: a Prospective Comparative Randomized Clinical Trial
Brief Title: Effectiveness of a Self-rehabilitation Program
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Centre Hospitalier Universitaire de Saint Etienne (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 1008155; 2010-A01369-30 (Other: ANSM)
Record Dates: First submitted 2015-09-11; First posted 2015-09-15 (Estimated); Last update posted 2017-01-18 (Estimated); Status verified 2017-01

CONDITIONS: Cervicalgia
Keywords: Cervicalgia; self-rehabilitation; physiotherapy
MeSH Terms: conditions — Neck Pain | interventions — Physical Therapy Modalities

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- self-rehabilitation + physiotherapy (Experimental): Patients will have, in addition to conventional physiotherapy, to visit two training sessions in self-rehabilitation at the hospital. They will then perform a self-rehabilitation / day session.
  Interventions: Other: self-rehabilitation + physiotherapy
- physiotherapy (Active Comparator): Patients will have only conventional physiotherapy
  Interventions: Other: physiotherapy

INTERVENTIONS:
Other: self-rehabilitation + physiotherapy — 2 training sessions in self-rehabilitation at the hospital and then a self-rehabilitation / day session + 14 physiotherapy sessions (2 by week)
  Arms: self-rehabilitation + physiotherapy
Other: physiotherapy — 14 physiotherapy sessions (2 by week)
  Arms: physiotherapy

SUMMARY:
The prevalence of non-specific neck pain is 12.1 / 1000 patients / year. Their support is most often based on analgesics combined with physical therapy. More recently authors have advocated the use of self-rehabilitation, that is to say, the use by the patient himself of physiotherapy exercises to perform at home regularly. However, if there are currently many studies on the effectiveness of self-rehabilitation for low back pain, there are few data on neck pain.

In this context we have chosen to implement a prospective, randomized study, on the effectiveness of self-rehabilitation in patients with chronic neck pain.

DETAILED DESCRIPTION:
Patients included in the "self-rehabilitation" group will, in addition to conventional physiotherapy, to visit two training sessions in self-rehabilitation at the hospital. Each patient received a booklet including advices to perform different kinds of exercises at home. The patients learn the exercises with the help of the physiotherapist and have to traine daily at home.

Patients will have to answer questionnaires about their pain at follow-usual consultations of their disease at 2 months and 4 months after the start physical therapy and during a phone call after 1 year.

ELIGIBILITY:
Inclusion Criteria:

* Non-specific neck pain * ≥ 15 days / month for more than 3 months
* Consultation first line in the pain center
* Subject able to complete questionnaires
* Subject able to understand and perform exercises

Exclusion Criteria:

* History of stroke
* History of carotid or vertebral arterial dissection
* "Whiplash" for less than six months
* Cervicobrachial neuralgia for less than 3 months
* Syndrome of thoracic outlet diagnosed
* Tumor and infectious syndromes
* Polyarthritis or major cervical spondylosis against known-indicating active mobilization of the cervical spine
* Unbound bone trauma
* Patients with cognitive impairment prevents proper application instructions

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 106 (Actual)
Dates: Start 2011-03; Primary Completion 2016-12 (Actual); Study Completion 2016-12 (Actual)

PRIMARY OUTCOMES:
Cervical pain | 2 months
  Verbal Scale Digital (EVN) cervical pain average 11 points (from 0-10) in the last week

SECONDARY OUTCOMES:
cervical pain | 1 year
  Verbal Scale Digital (EVN) cervical pain average 11 points (from 0-10) in the last week
cervical pain | 4 months
  Verbal Scale Digital (EVN) cervical pain average 11 points (from 0-10) in the last week

CONTACTS AND LOCATIONS:
Overall Officials: Christelle CREAC'H, MD, Principal Investigator — CHU de SAINT-ETIENNE
Locations (1):
- CHU de SAINT-ETIENNE, Saint-Etienne, France